CLINICAL TRIAL: NCT03592758
Title: Ultrasound in Evaluation of Difficult Airway Management Predictive Indexes
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Alessandri, Principal investigator, University of Roma La Sapienza
Other Study IDs: UEDAM
Record Dates: First submitted 2018-06-19; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Airway Complication of Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ultrasound assessment: all patient are evaluated by an ultrasound assessment before general anaesthesia

SUMMARY:
evaluate the efficacy of the ultrasound approach in predicting difficult mask ventilation in a heterogeneous population of patients undergoing general anesthesia.

DETAILED DESCRIPTION:
Preoperative ultrasound of the upper airway and detection of 5 ultrasound measurements:

Trachea-skin distance at the level of the thyroid isthmus; Trachea-skin distance at the jugular level Front commissure-skin distance; Distance from skin to the thyroid membrane Distance between hyoid bone and skin. Comparison of this measurement with HAN-scale for prediction of difficult mask ventilation during general anesthesia

ELIGIBILITY:
Inclusion Criteria:

- all patient > 18years old undergoing general anesthesia for elective surgery

Exclusion Criteria:

* Patients with fractures of the bones of the facial mass;
* Patients with laryngeal tumors
* Patients previously undergoing demolition of the larynx or neck;
* Tracheostomized patients;
* Pregnancy;
* Inter-incisive distance <3 cm;
* severely limited cervical mobility;
* Patients who are not given muscle relaxants
* Patient rejection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patient > 18 ys undergoing general anesthesia for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
ultrasound assessment | Ultrasound assessment will be performed 30 minutes before induction of general anaesthesia and the mask ventilation evaluation will be performed 3 minutes after induction with ''Han scale".
  the association between the ultrasound measurement and the difficulty of mask ventilation measured with the "Han scale". "Han scale" classify mask-ventilation in five grade of progressive difficulty: 0) mask ventilation did not attempt, 1) easy 2) difficult and requiring oral airway 3) very difficult requiring two practitioners 4) unable to mask ventilate.
  "Han scale" is the only grading scale available used routinely in anesthesiologic assessment of bag-mask ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Umberto I - UNiversità Sapienzadi Roma, Roma, Italy

REFERENCES:
- [Derived] Alessandri F, Antenucci G, Piervincenzi E, Buonopane C, Bellucci R, Andreoli C, Alunni Fegatelli D, Ranieri MV, Bilotta F. Ultrasound as a new tool in the assessment of airway difficulties: An observational study. Eur J Anaesthesiol. 2019 Jul;36(7):509-515. doi: 10.1097/EJA.0000000000000989. PMID 31742568